CLINICAL TRIAL: NCT00079482
Title: A Randomized, Open-Label Study of Oral CEP-701 Administered in Sequence With Standard Chemotherapy to Patients With Relapsed Acute Myeloid Leukemia (AML) Expressing FLT-3 Activating Mutations
Brief Title: Study of CEP-701 (Lestaurtinib) in Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C701a/204/ON/US; NCT00483340 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — lestaurtinib; Cytarabine; Mitoxantrone; Etoposide; Drug Therapy, Combination

ARMS (2):
- 1 (Active Comparator): Induction chemotherapy with or without sequential treatment with oral CEP-701 at 80 mg bid. For patients with duration of first CR of 1 to 6 months, the induction regimen will be MEC.
  Interventions: Drug: CEP-701; Drug: Mitozantrone, Etoposide, Cytarabine (combination Chemotherapy)
- 2 (Active Comparator): Induction chemotherapy with or without sequential treatment with oral CEP-701 at 80 mg bid. For patients with duration of first CR of more than 6 months to 24 months, the induction regimen will be HiDAC.
  Interventions: Drug: CEP-701; Drug: high-dose cytarabine

INTERVENTIONS:
Drug: CEP-701
  Other Names: lestaurtinib
Drug: high-dose cytarabine — Chemotherapy
  Other Names: HiDAC
  Arms: 2
Drug: Mitozantrone, Etoposide, Cytarabine (combination Chemotherapy) — Chemotherapy
  Other Names: MEC
  Arms: 1

SUMMARY:
The purpose of the study is to determine whether CEP-701 given in sequence with induction chemotherapy increases the proportion of patients with relapsed acute myeloid leukemia (AML) who achieve a second complete remission (CR).

DETAILED DESCRIPTION:
Patients randomly assigned to chemotherapy alone received the second course of induction chemotherapy as soon as clinically indicated; patients randomly assigned to receive chemotherapy plus sequential lestaurtinib had lestaurtinib withheld for 3 days (72 hours) before the start of the second 5-day course of chemotherapy and resumed lestaurtinib treatment 2 days (48 hours) after the final administration of the second course of chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* cytological confirmation of AML;
* relapsed disease following first CR of 1 month(30days)to 24 months(730days). The time from first relapse to study entry (start of first course of induction chemotherapy) must be no longer than 30days;
* confirmation of FLT-3 activating mutation positive status after point of initial relapse;
* aged 18 years or older;
* written informed consent;
* ability to understand and comply with study restrictions;
* no comorbid conditions that would limit life expectancy to less than 3 months;
* ECOG Performance Score of 0, 1,or 2;
* women must be neither pregnant nor lactating, and either of non-childbearing potential or using adequate contraception with a negative pregnancy test at study entry

Exclusion criteria:

* bilirubin > 2x ULN;
* ALT/AST > 3x ULN;
* serum creatinine > 1.5 mg/dL;
* resting ejection fraction of left ventricle l < 45%(applies only to patients scheduled to receive mitoxantrone, etoposide, and cytarabine [MEC];
* untreated or progressive infection;
* any physical or psychiatric cdtn that may compromise participation in the study;
* known CNS involvement with AML;
* any previous treatment with a FLT-3 inhibitor;
* requires current treatment for HIV with protease inhibitors;
* active GI ulceration or bleeding;
* use of an investigational drug that is not expected to be cleared by the start of CEP-701 treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2003-10; Primary Completion 2009-03 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine whether CEP-701 given in sequence with induction chemotherapy increases the proportion of patients with relapsed AML who achieve a second complete remission or a complete remission with incomplete platelet count recovery. | 113 days

SECONDARY OUTCOMES:
- overall survival - event-free survival - remission duration - safety and tolerability of CEP-701 - pharmacokinetics of CEP-701 - CEP-701 inhibitory activity | 113 days

CONTACTS AND LOCATIONS:
Locations (77):
- United States (34):
  - University of Alabama, Birmingham, Alabama
  - Mayo-Scottsdale, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Cancer Center, Los Angeles, California
  - Stanford Medical Center, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - ACORN-Central Georgia Hematology/Oncology, Macon, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - St. Francis Cancer Care Services, Beech Grove, Indiana
  - Indiana Cancer Pavillion, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - LSU Shreveport, Shreveport, Louisiana
  - Univeristy of Maryland Medicine - Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - Beth Israel Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Presbyterian, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - ACORN-The West Clinic, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
- Australia (7):
  - Call For Information, Sydney, New South Wales
  - Call for Information, Herston, Queensland
  - Call For Information, South Brisbane, Queensland
  - Call For Information, Adelaide, South Australia
  - Call For Information, Fitzroy, Victoria
  - Call For Information, Melbourne, Victoria
  - Call For Information, Perth, Western Australia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - CHA Hospital Enfant-Jesus, Québec, Quebec
- Germany (6):
  - Call For Information, Chemnitz
  - Call For Information, Dresden
  - Call For Information, Frankfurt
  - Call For Information, Heidelberg
  - Call For Information, Münster
  - Call For Information, Stuttgart
- Israel (3):
  - Call For Information, Haifa
  - Call For Information, Petah Tikva
  - Call For Information, Tel Litwinsky
- Italy (3):
  - Call For Information, Bologna
  - Call For Information, Roma
  - Call For Information, Turin
- Call For Information, Auckland, Auckland, New Zealand
- Poland (9):
  - Call For Information, Bialystok
  - Call For Information, Gdansk
  - Call For Information, Katowice
  - Call For Information, Krakow
  - Call For Information, Lodz
  - Call For Information, Lublin
  - Call For Information, Poznan
  - Call For Information, Warsaw
  - Call For Information, Wroclaw
- Romania (2):
  - Call For Information, Bucharest
  - Call For Information, Iași
- Russia (3):
  - Call For Information, Moscow
  - Call For Information, Novosibirsk
  - Call For Information, Saint Petersburg
- Spain (2):
  - Call For Information, Barcelona
  - Call For Information, Valencia
- Sweden (2):
  - Call For Information, Lund
  - Call For Information, Stockholm
- Ukraine (3):
  - Call For Information, Cherkassy
  - Call For Information, Kiev
  - Call For Information, Lviv

REFERENCES:
- [Derived] Levis M, Ravandi F, Wang ES, Baer MR, Perl A, Coutre S, Erba H, Stuart RK, Baccarani M, Cripe LD, Tallman MS, Meloni G, Godley LA, Langston AA, Amadori S, Lewis ID, Nagler A, Stone R, Yee K, Advani A, Douer D, Wiktor-Jedrzejczak W, Juliusson G, Litzow MR, Petersdorf S, Sanz M, Kantarjian HM, Sato T, Tremmel L, Bensen-Kennedy DM, Small D, Smith BD. Results from a randomized trial of salvage chemotherapy followed by lestaurtinib for patients with FLT3 mutant AML in first relapse. Blood. 2011 Mar 24;117(12):3294-301. doi: 10.1182/blood-2010-08-301796. Epub 2011 Jan 26. PMID 21270442